CLINICAL TRIAL: NCT04079309
Title: Anxiolytic Effects of Lavender and Orange Oil on Parents of Pediatric Patients With Dental Treatment Under Sedation
Brief Title: Anxiolytic Effects of Lavender and Orange Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cagil Vural, Lecturer, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09/05
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Anxiety State; Pediatric ALL; Dental Anxiety; Oil; Inhalation; Anesthesia
Keywords: Perioperative Anxiety; Lavender Oil; Orange Oil; Pediatric Dentistry; Deep Sedation
MeSH Terms: conditions — Anxiety Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Intervention (No Intervention): No mist will be diffused into the environment.
- Lavender (Active Comparator): 0,3 ml lavender oil diluted in 120 ml water will be diffused into the environment with (17-33 ml mist output per hour).
  Interventions: Behavioral: Lavender/Orange
- Orange (Active Comparator): 0,3 ml orange oil diluted in 120 ml water will be diffused into the environment with (17-33 ml mist output per hour).
  Interventions: Behavioral: Lavender/Orange

INTERVENTIONS:
Behavioral: Lavender/Orange — A diffuser containing 120 ml water and 0.3 ml lavender oil / 0.3 ml orange oil will be set into the parents' perioperative waiting rooms to mist at least 1 hour before the parent arrive.
  Arms: Lavender; Orange

SUMMARY:
The aim of this study is to determine the possible anxiety reducing effects of lavender oil and orange oil on parents with children receiving dental care under sedation during perioperative wait.

DETAILED DESCRIPTION:
Anxiety is a common problem for parents with children under sedation. It has long been known that operations, unconsciousness, the risks of the anesthesia and airway problems can cause a considerable amount of anxiety. Anxiety is associated with an uncertain psychological distress , and may vary to minor disturbances to extreme stress. The study aims to help parents improve their satisfaction by reducing their anxiety levels and ensure they have a better experience. In addition, anxiety can also prevent active participation of the parents during postoperative recovery. The physical and psychological effects of essential oils and traditional medicine practices as aromatherapy has been used for a long time and has potency to reduce using sedatives. Lavender oil is a fragrance that many of us have experienced in growing up at home and is also popular today. The lavender plant belongs to the Labitae family and has been used for centuries in dried or essential oil form. Lavender is obtained from flower heads and leaves with vapor distillation. This oil has also been specifically investigated and is an essential oil scientifically shown to reduce patient anxiety before various interventions. Orange oil is an essential oil produced by cells within the rind of an orange fruit (Citrus sinensis fruit). In contrast to most essential oils, it is extracted as a by-product of orange juice production by centrifugation, producing a cold-pressed oil. It is composed of mostly d-limonene. This oil has been investigated and shown to reduce anxiety and improve mood before various interventions.The anxiolytic effects of these essential oils has not been investigated for parents with children undergoing pediatric dental procedures under sedation.

The aim of this study is to investigate the effects of lavender oil and orange oil diffused in the perioperative waiting room of parents with children under sedation.

ELIGIBILITY:
Inclusion Criteria:

To be the parent of a child undergoing pediatric procedures under deep sedation.

To be over 18 years old. Volunteering to fill pre-operative anxiety tests.

Exclusion Criteria:

Hypersensitivity to lavender/orange and its products. Being on any medication. Being a psychiatric or psychological problem and being under treatment. Current upper airway infection or asthma story. Not want to be involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Reduction of preoperative anxiety | STAI will be applied at administration and after 1 hour waiting time.
  State Trait Anxiety Inventory (STAI) questionnaire will be applied. Turkish STAI consists of 2 questionnaires. The first survey measures state anxiety, while the second survey measures continuing anxiety(20 questions each).The STAI is a self-assessing and self-reporting anxiety questionnaire. The reliability and validity of the questionnaire are proven by numerous studies and the Turkish version is a reliable and valid questionnaire.
  All questions are rated on a 4-point scale (from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
  Internal consistency coefficients for the scale have ranged from .86 to .95; test-retest reliability coefficients have ranged from .65 to .75 over a 2-month interval (Spielberger et al., 1983). Test-retest coefficients for this measure in the present study ranged from .69 to .89. Considerable evidence attests to the construct and concurrent validity of the scale (Spielberger, 1989).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No